CLINICAL TRIAL: NCT01993628
Title: Constructional Apraxia in Alzheimer's Disease (AD) and Lewy Body's Dementia (LBD)
Brief Title: Construction-LBD (Constructional Apraxia in Alzheimer's Disease (AD) and Lewy Body's Dementia (LBD))
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 5565
Record Dates: First submitted 2013-10-31; First posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Alzheimer's Disease; Lewy Body's Dementia
MeSH Terms: conditions — Alzheimer Disease

ARMS (2):
- Alzheimer's disease (AD) (Experimental): Rey figure test and MRI
  Interventions: Other: Rey figure test; Other: MRI
- Lewy body's dementia (LBD) (Experimental): Rey figure test and MRI
  Interventions: Other: Rey figure test; Other: MRI

INTERVENTIONS:
Other: Rey figure test
Other: MRI

SUMMARY:
Alzheimer's disease (AD) and Lewy body's dementia (LBD) are two frequent neurodegenerative pathologies. They differ in their expression, their evolution but share same features which make their diagnosis uneasy.

Constructional apraxia has been described in both disease.The underlying mechanisms have been less studied and could be different in AD and LBD.

The definition of the constructional apraxia is purely descriptive and few models are inconclusive.

It is admitted that drawing tasks involve visuo-perceptive and visuo-spatial abilities, executive functions and working memory as well as purely "constructive" skills.

Regarding to different studies, visuo-perceptive abilities are more severely impaired in LBD than in AD and are considered as an early onset sign of the disease.

Executive functions deficits are documented in AD and LDB and could contribute to the drawing impairment.

It is possible to compensate the planning disorders in giving patient the best strategy to use.

If drawing impairment persists, they should result of others mechanisms like visuo-perception, visuo-spatial or constructive deficits.

The investigators suggest that giving the best planning strategy will help more AD patients who are supposed to fail in raison of an executive impairment, than the LDB group who is supposed to present visuo-perceptive deficits. An MRI will be proposed to study the cerebral areas involved in constructional apraxia.

ELIGIBILITY:
Inclusion Criteria:

* Alzheimer's disease or Lewy bodies dementia
* ≥ 45 years
* the cognitive impairment is mild to moderate
* French speaker
* a caregiver is present
* An informed consent is signed by the patient and the p.i.

Exclusion Criteria:

* MRI contraindication
* Other neurological disease (FTD, brain tumor, vascular disease…)
* Psychiatric disease (Schizophrenia, major depression, psychotic disorders, melancholia…)
* Patient who doesn't want to be informed in case of the discovery of an abnormality
* View or audition deficits, or motor disability which can interfere with the cognitive testing
* Patient participating to an exclusive protocol or in the period of exclusion
* Pregnant woman
* Person under an administrative or legal measure of liberty privation
* Person under a legal measure of protection or under administrative supervision
* Person unable to give his consent

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2013-10; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Score obtained at the Rey figure test with a planning strategy help by LBD patients compared to the score obtained by AD patients. | At inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France